CLINICAL TRIAL: NCT07219056
Title: The Effect of the Safe and Sound Protocol on Emotional Regulation in Traumatized Adults With Substance Use Disorders
Brief Title: Safe & Sound Protocol in Adults With Trauma and SUD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Caron Treatment Centers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Caron002
Record Dates: First submitted 2025-10-14; First posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Substance Use Disorders; Posttraumatic Stress Symptom; Anxiety
Keywords: substance use disorders; posttraumatic stress symptoms; anxiety
MeSH Terms: conditions — Substance-Related Disorders; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This is a two-armed, prospective, randomized, double-blind, sham-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, all study staff including the PI, and clinical staff will be blinded to the group assignment. The PI will remain unblinded as they created the randomization design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active SSP (Experimental): Participants will engage with the SSP for a minimum of 3 hours and a maximum of 5 hours over the course of seven days.
  Interventions: Device: Safe and Sound Protocol
- Sham SSP (Sham Comparator): Participants will engage with the SSP for a minimum of 3 hours and a maximum of 5 hours over the course of seven days. The sham protocol will deliver unfiltered music.
  Interventions: Device: Safe and Sound Protocol

INTERVENTIONS:
Device: Safe and Sound Protocol — Participants will complete a series of instruments after consenting to participate and have the SSP uploaded onto their mobile device or tablet. Participants will listen to the SSP for 3 to 5 hours over the course of 7 days. On the eighth day, participants will complete a follow-up set of instruments. The active arm will deliver the actual SSP intervention whereas the sham arm will deliver unfiltered music.
  Other Names: SSP

SUMMARY:
This study will explore whether the use of the Safe and Sound Protocol (SSP) app is an effective adjunct to treatment as usual (TAU) in individuals with co-occurring substance use disorders and trauma. This study will recruit 129 participants (100 completers) randomized to receive either active or sham SSP in addition to TAU. Participants will utilize the SSP for a minimum of three hours to a maximum of five hours for a total of seven days. Data will be collected at both pre- and post-test. Data to be collected will include measures on affect, anxiety, personality, mindfulness, and posttraumatic stress disorder symptoms. The SSP has shown effectiveness in reducing symptoms of anxiety, depression, and trauma symptoms in pilot studies conducted at other locations. This will be the first study to examine the effectiveness of SSP with individuals with co-occurring SUD and trauma.

DETAILED DESCRIPTION:
The Safe and Sound Protocol (SSP) was developed by Dr. Stephen Porges based on his Polyvagal Theory that highlights the vagus nerve's influences on emotional and behavioral regulation, social connection, and fear/trauma responses.

Research examining the effectiveness of SSP with children and/or adults on the Autism Spectrum has shown improvement in social awareness and decline in auditory hypersensitivities and hypo-sensitivities, visual sensitivity, tactile hypersensitivities, selective eating and digestive problems. SSP has also been shown to reduce symptoms of anxiety, depression and autonomic reactivity in individuals engaged in speech therapy for voice and throat complaints.

There is on-going clinical research to examine the effectiveness of SSP in various populations, including those suffering from posttraumatic stress disorder (PTSD). In real-world data obtain through the SSP platform, just over half of individuals reporting clinical levels of PTSD symptoms as assessed on the Posttraumatic Checklist - 5 (PCL-5) had a reduction in symptoms to below the clinical threshold following the completion of SSP.

Safe and Sound Protocol (SSP) Core is five hours of music therapy that is progressively filtered through a patented algorithm that highlights middle sound frequencies, the frequency most associated with cues of safety from human speech. This is designed to stimulate the vagus nerve by engaging the middle ear muscles and nerves to move out of defensive state of activation and activate the social engagement and calming system of the nervous system. SSP is designed to help participants regulate their nervous system to support reduction in distress and increased social connection.

To date, there is no research underway to examine the effectiveness of SSP for individuals experiencing posttraumatic stress symptoms and a substance use disorder (SUD). Individuals experiencing posttraumatic stress symptoms and SUD are hypothesized to benefit from a non-invasive treatment designed to regulate their autonomic nervous system, such as SSP.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 years old to 75 years old
* In residential treatment for substance use disorder.
* Has a history of trauma and is enrolled in Caron's trauma programming
* Is proficient in English
* Able to provide written informed consent.
* Stated willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

* Does not speak English
* Age < 18 or > 75
* Does not have a history of trauma
* Active psychosis
* Active or uncontrolled seizures
* Tinnitus
* Active suicidal ideation
* Actively engaging in self-injurious behavior
* Severe neurological condition
* Diagnosis of autism
* Has any serious medical disease or mental health condition which, in the judgment of the Principal Investigator or his/her designee, would make study participation unsafe, or would make intervention compliance difficult.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Difference in posttraumatic stress symptom scores pre-post between groups as measured by the Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5). | Day 1 and Day 8
  Linear mixed effects models for repeated measurements will be used to evaluate the difference in changes in posttraumatic stress symptom outcomes between treatment and sham group.
Difference in anxiety symptom scores pre-post between groups as measured by the Generalized Anxiety Disorder-7 (GAD-7) scale. | Day 1 and Day 8
  Linear mixed effects models for repeated measurements will be used to evaluate the difference in changes in anxiety outcomes between treatment and sham group.
Difference in autonomic arousal symptom scores pre-post between groups as measured by the Body Perception Questionnaire Autonomic Symptoms - short form (BPQ-20 ANS). | Day 1 and Day 8
  Linear mixed effects models for repeated measurements will be used to evaluate the difference in changes autonomic arousal outcomes between treatment and sham group.

SECONDARY OUTCOMES:
Differences in positive and negative affect scores pre-post between groups as measured by the Positive and Negative Affect Schedule. | Day 1 and Day 8
  Linear mixed effects models for repeated measurements will be used to evaluate the difference in changes in positive and negative affect outcomes between treatment and sham group.
Changes in mindfulness scores pre-post between groups as measured by the Cognitive and Affective Mindfulness Scale - Revised (CAMS-R) | Day 1 and Day 8
  Linear mixed effects models for repeated measurements will be used to evaluate the difference in changes in mindfulness outcomes between treatment and sham group.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Deneke, PhD, Principal Investigator — Caron Treatment Centers
Locations (1):
- Caron Treatment Centers, Wernersville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared